CLINICAL TRIAL: NCT02637180
Title: A Multiple Center, Prospective Study Targeting the Secondary Prevention of Fractures in Greece: Evaluation of the Fracture Liaison Service in Multiple Hospital Settings
Brief Title: Secondary Prevention of Osteoporotic Fractures: a Multiple Center Fracture Liaison Service in Greece
Status: Completed | Type: Observational
Sponsor: Hellenic Society for the Study of Bone Metabolism (Other)
Collaborators: Democritus University of Thrace (Other); Aristotle University Of Thessaloniki (Other); UNIVERSITY OF THESSALIA, SCHOOL OF HEALTH SCIENCES (Unknown); National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: EEMMO/FLS/2015
Record Dates: First submitted 2015-12-12; First posted 2015-12-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Osteoporosis
Keywords: osteoporosis; fracture; liaison service
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with low-energy fracture(s): The study will include patients from pre-defined groups of individuals (postmenopausal, perimenopausal, male, and steroid induced osteoporosis) who would be anyway eligible to receive treatment for their condition according to standard medical practice and Greek treatment guidelines.
  Drug: anti-osteoporotic medication (bisphosphonates, denosumab, strontium ranelate, teriparatide, SERMs)
  Interventions: Drug: anti-osteoporotic medication

INTERVENTIONS:
Drug: anti-osteoporotic medication — check previous information
  Other Names: all available anti-osteoporotic medication

SUMMARY:
This is multiple center, prospective study aiming to investigate the tracking and outcome of patients attending Greek General hospitals with low-trauma fractures. Secondary end-points were to facilitate the implementation of coordinated, multi-disciplinary models of care for secondary fracture prevention, and to monitor osteoporosis treatment initiation, osteoporosis treatment persistence at 12 months, compliance, and subsequent fractures.

DETAILED DESCRIPTION:
This study includes 5 different hospitals in 4 cities of Greece. The responsible party in each hospital is an orthopedic department which will organize a fracture liaison service (FLS) for both Hospitalized patients over 50 years old with low energy fractures and Outpatients over 50 years old with low energy fractures (low energy fracture is defined as a fracture resulting from minimal trauma such as falling from standing height or less).

This action targets to improve patient care and to reduce secondary osteoporotic fractures, along with collateral healthcare cost.

Prerequisite for patients' enrollment in the FLS program is the voluntary signed acceptance of the program's terms and conditions (signed Inform Consent Forms).

Program Services for eligible patients include the following steps:

* The FLS personnel informs patient about the program, its services and provides him/her with the relevant, informative, printed material. After obtaining patient's signed informed consent, the competent personnel in cooperation with treating physicians:

  1. Compiles and updates patient's file.
  2. Ensures that diagnostics and laboratory tests will include: Hip and Lumbar Spine BMD (of at least one hip, in two points of lumbar spine if possible); Thoracic Spine F/P & Lumbar Spine F/P X-rays; and the minimum required laboratory test for patients with low energy fracture, that are candidates to receive "anti-osteoporotic" medication, according to Greek osteoporosis guidelines. Calculates the relevant FRAX score.

  3) Assures that treating physician (or the physician accountable for the bone metabolic disorders) recommends a treatment for the prevention of a new fracture, if appropriate, after patient's examination and before patient leaves hospital.
* The FLS personnel ensures the restoration of regular contact with the fractured patients, aiming to inform and alert them (and/or their relatives, families), by reminding and facilitating the next appointment in outpatient office for Metabolic Bone Diseases.
* The FLS personnel compiles and applies a patient support program, with regular telephone contacts. The program informs, awares, motivates and facilitates patients to follow up with a specialized physician, by providing useful information or/and services (for example: to schedule the next appointment in the specific hospital's outpatient office). During the telephone contact specific data will be collected and recorded, such as if a new fracture has emerged, if patient is under regular supervision / follow up by physician for osteoporosis, if patient is still under treatment. If not the discontinuation reason should be collected. The telephone contact schedule will be as follows: One, six and twelve months after discharge from hospital.

The enrollment period lasts 365 days in each hospital, starting from first patient's enrollment date in each particular center. Patients' follow up will also last 365 days and therefore the total duration of the program is 2 years in every center.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients and Outpatients over 50 years old with low energy fractures (low energy fracture is defined as a fracture resulting from minimal trauma such as falling from standing height or less).

Exclusion Criteria:

* Presence of osteomalacia and/or other clinical entities predisposing to low energy fractures, apart from osteoporosis, such as primary or secondary hyperparathyroidism, Paget's disease of bone, osteogenesis imperfecta and paraplegia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 50 years old with low energy fractures
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Participation rate in the FLS program | 2 years
  Participation rate in the FLS program of patients with low-trauma fractures

SECONDARY OUTCOMES:
Percentage of patients initiating osteoporosis treatment | 2 years
percentage of patients experiencing subsequent fractures | 2 years
osteoporosis treatment adherence at 24 months [measured by Medication Possession Ratio (MPR)] | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christos Kosmidis, MD, Phd, Principal Investigator — Hellenic Society for the Study of Bone Metabolism
Locations (4):
- Greece (4):
  - NATIONAL AND KAPODISTRIAN UNIVERSITY OF ATHENS, MEDICAL SCHOOL, 2nd DEPARTMENT OF ORTHOPAEDIC SURGERY, Athens, Attica
  - Democritus University of Thrace, School of Medicine, Department of Orthopaedic Surgery, Alexandroupoli, Evros
  - Orthopaedic Department, Faculty of Medicine, School of Health Sciences, University of Thessalia, Larissa
  - Aristotle University of Thessaloniki, 3rd University Orthopaedic Department, Papageorgiou General Hospital, Thessaloniki

REFERENCES:
- [Background] Marsh D, Akesson K, Beaton DE, Bogoch ER, Boonen S, Brandi ML, McLellan AR, Mitchell PJ, Sale JE, Wahl DA; IOF CSA Fracture Working Group. Coordinator-based systems for secondary prevention in fragility fracture patients. Osteoporos Int. 2011 Jul;22(7):2051-65. doi: 10.1007/s00198-011-1642-x. Epub 2011 May 24. PMID 21607807
- [Background] McLellan AR, Gallacher SJ, Fraser M, McQuillian C. The fracture liaison service: success of a program for the evaluation and management of patients with osteoporotic fracture. Osteoporos Int. 2003 Dec;14(12):1028-34. doi: 10.1007/s00198-003-1507-z. Epub 2003 Nov 5. PMID 14600804
- [Background] Cooper MS, Palmer AJ, Seibel MJ. Cost-effectiveness of the Concord Minimal Trauma Fracture Liaison service, a prospective, controlled fracture prevention study. Osteoporos Int. 2012 Jan;23(1):97-107. doi: 10.1007/s00198-011-1802-z. Epub 2011 Sep 28. PMID 21953475
- [Background] Makras P, Vaiopoulos G, Lyritis GP; Greek National Medicine Agency. 2011 guidelines for the diagnosis and treatment of osteoporosis in Greece. J Musculoskelet Neuronal Interact. 2012 Mar;12(1):38-42. No abstract available. PMID 22373950
- [Background] Dehamchia-Rehailia N, Ursu D, Henry-Desailly I, Fardellone P, Paccou J. Secondary prevention of osteoporotic fractures: evaluation of the Amiens University Hospital's fracture liaison service between January 2010 and December 2011. Osteoporos Int. 2014 Oct;25(10):2409-16. doi: 10.1007/s00198-014-2774-6. Epub 2014 Jul 1. PMID 24980182